CLINICAL TRIAL: NCT01805089
Title: A Randomized Trial of Oral Melatonin Supplementation in Breast Cancer Survivors
Brief Title: Melatonin Versus Placebo in Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Wendy Chen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-305
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin 3 mg (Active Comparator): Taken orally, once per day, at/around 9:00pm
  Interventions: Drug: Melatonin 3 mg
- Placebo (Placebo Comparator): Taken orally, once per day, at/around 9:00pm
  Interventions: Drug: Melatonin 3 mg

INTERVENTIONS:
Drug: Melatonin 3 mg — Melatonin vs. Placebo
  Other Names: Melatonin

SUMMARY:
The purpose of this research study is to determine whether melatonin taken every night can affect blood levels of estrogen or IGF (insulin-growth factor levels). Both IGF and estrogen are normally produced in the body and may influence breast cancer risk. Melatonin is also naturally produced in the body. Laboratory studies have shown that melatonin may decrease cancer growth and influence estrogen and IGF levels. Melatonin's effects on sleep, hot flashes, and mood will also be measured.

DETAILED DESCRIPTION:
If you agree to participate in this study you will be asked to undergo a blood test to find out if you are eligible. Approximately 2 tablespoons of blood will be drawn. The blood test will check your health and menopausal status. This test will aslo be used to help measure any additional effects of the study drug on your body. If you have had a blood test recently, it may or may not have to be repeated. If these tests show that you are eligible to participate in the research study, you will begin the study. If you do not meet the eligibility criteria, you will not be able to participate.

Because no one knows which of the study options is best, and all of the options are considered likely to work, you will be "randomized" into one of the study groups: melatonin or placebo.

Randomization means that you are put into a group by chance. It is like flipping a coin. Neither you nor the research doctor will choose what group you will be in. You will have an equal chance of being placed in either group. Neither you nor the research doctor will know what group you are in. You will not know the identity of your study treatment until after the final research analysis has taken place. Once this has happened, you will be mailed a letter from the principal research doctor telling you which study drug you received while on study.

You will be given a study drug and it will either contain melatonin or placebo (pills with no medical effect). You will take one tablet by mouth every night as close to 9:00 pm as possible. You should not make up missed doses. You will be given enough study drug to last 4 months. You will also be given a study medication-dosing calendar to write down times you took the study drug for each month you are taking the study drug.

Before taking the study drug, you will have blood tests to look at the level of estrogen and IGF in your blood. Approximately 2 tablespoons of blood will be drawn. At this visit, you will also be asked to complete a questionnaire that will take approximately 15 minutes.

A member of the research study staff will check in by telephone once a month to monitor your experiences on the research study. You may also contact a member of the research study staff at any time if you have any questions or concerns.

You should tell your research doctor if you are currently taking black cohosh, flaxseed or soy in pill or supplement form, as it may affect your participation in this research study.

After you have completed approximately 4 months of study drug, you will return to clinic to see a member of the research study staff. At this visit you will have the following tests and procedures: You will have blood tests to look at the level of estrogen and IGF in your blood. Approximately 2 tablespoons of blood will be drawn. You must return your study medication-dosing calendar and all of your pill bottles at the end of the research study to a member of the research study staff. You wil also be asked to complete a questionnaire that will take about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* History of ductal carcinoma in situ, lobular carcinoma in situ or stages 1-3 breast cancer
* Not currently receiving chemotherapy or hormonal therapy
* Postmenopausal

Exclusion Criteria:

* Stage IV breast cancer or systemic recurrences
* Prior malignancies of any type other than breast cancer, basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Use of adjuvant hormonal therapy, oral estrogen or progesterone replacement therapy, lutenizing hormone releasing hormone agonists currently or within the past 60 days
* Concomitant use of beta-blockers
* Concomitant nightly use of sleep aids at bedtime
* Working more than one overnight shift per month on a regular basis
* Concomitant use of postmenopausal hormone replacement therapy
* Concomitant use of black cohosh, flaxseed or soy in pill or supplement form
* Use of any type of oral melatonin supplementation within the past 30 days
* Use of warfarin (coumadin) within the past 30 days
* Active seizure disorder requiring the use of daily anti-epileptic medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Chen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Melatonin 3mg: Taken orally, once per day, at/around 9:00pm
  Melatonin
- Placebo: Taken orally, once per day, at/around 9:00pm
  Placebo
Period: Overall Study
Arm/Group | Melatonin 3mg | Placebo
Started | 48 | 47
Completed | 43 | 43
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Melatonin: Taken orally, once per day, at/around 9:00pm
  Melatonin
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Median (Full Range); unit: years] | 58 [48 to 70] | 60 [38 to 71] | 59 [38 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 95
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 46 | 45 | 91
  African American | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Multi-racial | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 47 | 95
Cancer Stage [Number; unit: participants]
  Stage 0 | 6 | 6 | 12
  Stage I | 21 | 15 | 36
  Stage II | 15 | 22 | 37
  Stage III | 6 | 4 | 10
Smoking Status [Number; unit: participants]
  Missing | 0 | 1 | 1
  Current Smoker | 1 | 1 | 2
  Non-Smoker | 25 | 22 | 47
  Former Smoker | 22 | 23 | 45
Body Mass Index (BMI) [Median (Full Range); unit: Kg/m2] | 25.7 [20.1 to 44.9] | 25.0 [19.1 to 39.6] | 25.6 [19.1 to 44.9]
Estradiol [Mean (Standard Deviation); unit: pg/ml] | 4.59 (4.03) | 3.35 (2.19) | 3.97 (3.29)
Insulin-like Growth Factor 1 [Mean (Standard Deviation); unit: ng/ml] | 181.95 (60.22) | 177.83 (46.67) | 179.89 (53.6)
Sleep (Pittsburgh Sleep Quality Index) [Mean (Standard Deviation); unit: units on a scale] — Pittsburgh Sleep Quality Index measures average sleep quality based on self-report over past 7 days. Range is 0 to 21. Higher values are considered worse. There are 7 subscales which are added together.
  units on a scale | 7.2 (4.2) | 5.5 (3.3) | 6.4 (3.9)
Hot Flashes [Mean (Standard Deviation); unit: hot flash score] | 5.5 (6.5) | 4.5 (5.2) | 5.1 (5.9)
Mood [Mean (Standard Deviation); unit: CESD global score] | 6.7 (5.5) | 6.0 (6.3) | 6.3 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Plasma Estradiol Levels After 4 Month Course of Melatonin or Placebo
Description: Absolute plasma estradiol levels after 4 month course of melatonin or placebo, only 4 month level provided below.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 43 | 43
pg/ml | 4.59 (3.42) | 3.39 (2.25)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Compliance
Description: To evaluate compliance with a 4 month course of melatonin. Compliance was assessed via pill counts.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 48 | 47
participants | 43 | 43

3. Secondary Outcome: Change in Mood, Sleep Quality and Menopausal Symptoms From Baseline to 4 Months
Description: Mood was assessed by the Center for Epidemiologic studies Depression Scale. The scale measures depressive symptoms in 20 items. Each question has a 4 point answer (0-3) so the scale range is 0-60. A higher score indicates more depression. Sleep quality was assessed by the Pittsburgh Sleep Quality Index. There are 19 questions each with a 3 point answer. The questions are grouped into 7 subscales and each has a value from 0-3. The 7 subscales are then added together to yield a global score with a range of 0-21. Higher scores indicate worse sleep. Menopausal symptoms were assessed by NCCTG Hot Flash diary. Subjects track the number and severity of hot flashes daily for 1 week. Subjects grade the severity of the hot flashes on a scale of 1-4, with 1 being mild and 4 very severe. Frequency and the severity determine the score . The minimum score is 0 (no hot flashes) and there is no maximum score. A higher score indicates more severe hot flashes. There are no subscales or no units.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: change in PSQI score
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 43 | 43
change in PSQI score
  Change in PSQI | -1.9 (2.4) | -0.1 (2.0)
  Change in CESD | -0.2 (4.6) | -0.0 (5.4)
  Change in Hot Flash Score | -1.0 (6.1) | -1.3 (3.9)

ADVERSE EVENTS:
Time Frame: During 4 months of study treatment
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 7/48 | 1/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=48) | Placebo (N=47)
Headache (Nervous system disorders) | 3 | 0
Bad Dreams (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No